CLINICAL TRIAL: NCT00151684
Title: Diazoxide-Mediated Insulin Suppression in Hyperinsulinemic Obese Men: a Dose Response Study, Part II
Brief Title: Diazoxide-Mediated Insulin Suppression in Hyperinsulinemic Obese Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTC-268-060504
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2008-02

CONDITIONS: Obesity; Hyperinsulinism
Keywords: Obesity; Hyperinsulinism; Diazoxide
MeSH Terms: conditions — Obesity; Hyperinsulinism | interventions — Diazoxide

INTERVENTIONS:
Drug: Diazoxide

SUMMARY:
The purpose of this study is to explore diazoxide efficacy in treatment of obese men and assessment of maximal insulin suppression in obese men without hyperglycaemia.

Obesity is associated with markedly elevated plasma insulin levels throughout the day. The concept is that obese subjects predominantly develop lean tissue resistance against the glucoregulatory actions of insulin, but remain relatively sensitive to the lipogenic and antilipolytic effects of insulin in adipose tissue. According to this theory, suppression of hyperinsulinism by diazoxide, a well known inhibitor of glucose stimulated insulin secretion, might be useful to treat obesity because it will help to reverse the process of lipid storage.

DETAILED DESCRIPTION:
The purpose of this study is to explore diazoxide efficacy in treatment of obese men and assessment of maximal insulin suppression in obese men without hyperglycaemia.

Study design:

This study is an open-labelled, non-randomized, phase IIa study.

Treatment:

During a 6 month period, the dosage of Diazoxide will be raised gradually until a maximum of 900 mg/day, under control of bloodpressure and glucose levels.

Endpoints, monthly determined:

* body weight
* abdominal circumference
* body composition measured by Dual Energy X-ray Absorptiometry
* glucose tolerance

ELIGIBILITY:
Inclusion Criteria:

* fasting glucose < 7.0 mmol/L
* fasting C-peptide plasma level > 1.0 nmol/L
* HbA1c of 6.0% or lower
* Absence of comorbidity
* Absence of medication use

Exclusion Criteria:

* Plasma Creatinine > 120 micromol/L
* Liverenzymes > 2 times the upper normal limit
* Gout
* Alcohol use > 2 units/day
* Illicit drug use
* Quit smoking less than 6 months ago

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2004-11

PRIMARY OUTCOMES:
body weight
abdominal circumference
body composition measured by Dual Energy X-ray Absorptiometry
glucose tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Hans de Boer, MD PhD, Principal Investigator — Rijnstate Hospital, Arnhem, The Netherlands
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands

REFERENCES:
- [Background] Schreuder T, Karreman M, Rennings A, Ruinemans-Koerts J, Jansen M, de Boer H. Diazoxide-mediated insulin suppression in obese men: a dose-response study. Diabetes Obes Metab. 2005 May;7(3):239-45. doi: 10.1111/j.1463-1326.2004.00449.x. PMID 15811140